CLINICAL TRIAL: NCT00483275
Title: Effects of a Multi-modal 12-month-intervention With Alfacalcidol Plus Calcium, Patient Education and a Mobility Program on the Number of Fallers Among Patients With an Impaired Kidney Function Aged 65 and Older.
Brief Title: Fall Prevention by Alfacalcidol and Training
Acronym: SPALT
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: No final agreement with sponsor
Sponsor: Ruhr University of Bochum (Other)
Collaborators: Teva Branded Pharmaceutical Products R&D, Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: GER-001-SP; EudraCT 2006-006205-83
Record Dates: First submitted 2007-06-06; First posted 2007-06-07 (Estimated); Last update posted 2011-07-21 (Estimated); Status verified 2011-07

CONDITIONS: Accidental Falls; Chronic Renal Insufficiency; Aged
Keywords: Accidental Falls; Accident Prevention; Patient Education; Exercise Training; Alfacalcidol
MeSH Terms: conditions — Renal Insufficiency, Chronic | interventions — alfacalcidol; Gait; Resistance Training; Patient Education as Topic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Alfacalcidol
Behavioral: Balance, gait and strength training
Behavioral: Patient education

SUMMARY:
Objective of the study is to evaluate the effect of a multimodal therapy on the basis of current guidelines on fall prevention consisting of a 12-months intervention with Alfacalcidol and calcium, patient education and a mobility program in a group of patients 65 years of age or older with an impaired renal function in comparison to a group receiving usual care.

DETAILED DESCRIPTION:
The risk of falling increases with age. An impaired renal function is an additional risk factor. Guidelines and systematic reviews suggest, that multimodal interventions are most likely to control this risk. This study evaluates, if patients at high risk for falls will benefit from a multimodal intervention simple and feasible enough to be transferred into general practice. Participants will be randomized either into an intervention group or a control group receiving usual care.

The multimodal intervention consists of:

* medication: Participants receive 1µg Alfacalcidol and 500mg Calcium daily
* mobility program: strength, balance and gait training twice a week for one hour
* patient education: a single meeting with teaching lessons on risk factors for falling and modes of fall prevention followed by an evaluation of the individual fall risk and corresponding recommendations to reduce it

ELIGIBILITY:
Inclusion Criteria:

* Men and women who are 65 years of age or older
* Personal history of at least one movement-related, non-syncopal fall, either within the past year OR earlier with additional findings of an increased fall risk during screening examination.
* Creatinine-clearance of 30 to 60 ml/min equivalent to a moderately impaired kidney function (stage 3) according to the classification of the Kidney Disease Outcomes Quality Initiative (K/DOQI) of the National Kidney Foundation (NKF).

Exclusion Criteria:

* Immobility with inability to go out and participate in training course
* History of a fracture or of a stroke provided the event has occurred in the last 3 months
* Presence of a physical or mental disorder that has led to a set-up or to a planned set-up for a statutory care
* Severe dementia
* Severe disorder of speech or comprehension
* Disease that rules out participation during the intervention period or that would deteriorate as a result of type of intervention (e.g. absorptive hypercalciuria, nephrocalcinosis, calcium containing renal calculi or hypophosphataemia)
* Hypersensitivity (allergy) to Alfacalcidol, groundnuts, groundnut oil or Soya
* Vitamin-D hypersensitivity or -intoxication
* Simultaneous intake of vitamin D and its derivatives.
* Participation in any other clinical trial, that is still ongoing or has been completed less than 3 months prior date of intended inclusion
* Substitution of more than 500 mg calcium per day
* Planned medical therapy during the period of intervention that requires long-term suspension of intervention.
* Presence of hypercapnia of over 2.6mmol/l, calcium x phosphate product of over 3.7 (mmol/l)2 and alkalosis with venous blood-pH- reading of over 7.44 (milk-alkali-syndrome, Burnett syndrome)
* Hypercalcaemia (e.g. as a result of hyperparathyroidism, an overdose of vitamin D, paraneoplastic syndrome, osseous metastases, sarcoidosis, Boeck´s disease, osteoporosis induced by immobilisation) or hypermagnesemia according to normative values of the engaged laboratory
* Hereditary fructose intolerance
* Commitment into an institution

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 484 (Estimated)
Dates: Start 2007-06; Study Completion 2009-09 (Estimated)

PRIMARY OUTCOMES:
Number of fallers | One year

SECONDARY OUTCOMES:
Number of falls | One year
Number of fractures | One year
Performance in balance and mobility | One year
Fear of falling | One year
Rate of hypercalcaemia | One year

CONTACTS AND LOCATIONS:
Overall Officials: Prof. Dr. med. Ludger Pientka, MD, MPH, Principal Investigator — Klinik für Altersmedizin und Frührehabilitation, Marienhospital Herne, Ruhr-Universität Bochum
Locations (1):
- Klinik für Altersmedizin und Frührehabilitation, Marienhospital, Ruhr-Universität Bochum, Herne, North Rhine-Westphalia, Germany